CLINICAL TRIAL: NCT06808451
Title: Diagnosis and Treatment of Urinary Tract Infection Using DNA PCR Versus Urine Culture - A Randomized Controlled Trial
Brief Title: Diagnosis and Treatment of Urinary Tract Infection Using DNA Polymerase Chain Reaction Versus Urine Culture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, David Sheyn, Director, Division of Urogynecology and Reconstructive Pelvic Surgery, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY20241345
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Urinary Tract Infections
Keywords: urine culture; DNA PCR
MeSH Terms: conditions — Urinary Tract Infections | interventions — Random Amplified Polymorphic DNA Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DNA Polymerase Chain Reaction (PCR) (Experimental): Gene analysis with PCR will be conducted from the urine samples of the patients with acute UTI symptoms.
  Interventions: Device: DNA PCR
- Urine Culture (Active Comparator): Urine samples of the patients with acute UTI symptoms will be sent to the UH lab for routine urine culture.
  Interventions: Diagnostic Test: Urine Culture

INTERVENTIONS:
Device: DNA PCR — Gene analysis with PCR will be conducted from the urine samples of the patients with acute UTI symptoms.
  Arms: DNA Polymerase Chain Reaction (PCR)
Diagnostic Test: Urine Culture — Urine samples of the patients with acute UTI symptoms will be sent to the UH lab for routine urine culture.
  Arms: Urine Culture

SUMMARY:
Adults 18 years or older with urinary tract infection (UTI) symptoms. Participants will be assigned to either the urine culture group or the DNA PCR study group by randomization. At time of enrollment in the study they will be also asked to fill out two questionnaires. If prescribed antibiotics for treatment of a UTI, participants will then be called the day after they are scheduled to stop their antibiotics. Participants will be asked to fill out questionnaires the day after finishing antibiotics. Participants will be enrolled in the study for a maximum of 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women 18 years and older
* Presenting to clinic with symptoms of UTI or cystitis
* Patients with Medicare and Medicaid insurance

Exclusion Criteria:

* Urinary diversion of any type
* Chronic indwelling urinary catheter
* Diagnosed UTI within the previous 21 days
* Antibiotic therapy within the previous 21 days
* Use of phenazopyridine within the previous 21 days
* Commercial insurance
* Non-English speaking
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms as measured by UTI-SIQ-8 questionnaire | Baseline, one day after antibiotic completion
  The UTI-SIQ-8 is an eight item questionnaire that asks about symptom severity and symptom impairment on a likert scale from 0 to 4, 0 being not at all and 4 being very strong/very severe.
Change in symptoms as measured by the UTI Symptom Assessment questionnaire | Baseline, one day after antibiotic completion
  The UTI Symptom Assessment questionnaire is a ten item questionnaire that asks about symptom relief, with lower scores indicating less symptoms.

SECONDARY OUTCOMES:
Length of time from patient presentation to initiation of treatment as measured by medical record review | Up to 21 days
Number of antibiotic changes as measured by medical record review | Up to 21 days
Duration of antibiotic use as measured by medical record review | Up to 21 days
  Duration will be measured in days
Number of times participant represents with UTI symptoms as measured by medical record review | Up to 30 days
  Duration will be measured in days
Number of additional diagnostic procedures related to initial presenting symptoms as measured by medical record review | Up to 21 days
Number of hospitalizations related to UTI as measured by medical record review | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: David Sheyn, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No